CLINICAL TRIAL: NCT00460135
Title: The Impact of Resistance Exercise Training On Metabolic Dysregulation in Obese Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Laurent Legault,MD, MUHC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PED-06-004
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Childhood Obesity; Body Composition; Resistance Training; Insulin Resistance
Keywords: Resistance; Training; Obesity; Children
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT (Experimental): resistance training
  Interventions: Behavioral: resistance training
- Routine care (No Intervention): General counseling on increasing physical exercise

INTERVENTIONS:
Behavioral: resistance training — 2 times a week resistance training
  Arms: RT

SUMMARY:
Impact of resistance training in prepubertal children with obesity focusing mostly in changes in body composition and markers of insulin resistance.

Hypothesis is that this will show positive changes in this randomized controlled trial.

DETAILED DESCRIPTION:
24 obese prepubertal obese children randomized to either resistance training program or usual care for 12 weeks. Baseline blood profiles and DEXA scans done before and after 12 weeks of training with the help of kinesiology graduates from Concordia University kinesiology department.

ELIGIBILITY:
Inclusion Criteria:

* Between 8-12y
* Prepubertal
* Not on medications with known impact on weight loss

Exclusion Criteria:

* Pubertal
* Uncontrolled thyroid condition
* Type 2 diabetes

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Changes in body composition as per DEXA scans | 12 weeks

SECONDARY OUTCOMES:
Changes in insulin resistance as per HOMA score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Legault, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada